CLINICAL TRIAL: NCT04388722
Title: Monitoring Noninvasively for Infusion and Transfusion Optimization in a Randomized (MONITOR) Trial
Brief Title: Monitoring Noninvasively for Infusion and Transfusion Optimization
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's decision to withdraw study.
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MONITOR
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Post Operative Hemorrhage; Transfusion Related Complication; Blood Transfusion Associated Adverse Reactions; Hypovolemia
MeSH Terms: conditions — Postoperative Hemorrhage; Transfusion Reaction; Hypovolemia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Arm (No Intervention)
- Investigational Arm (Experimental)
  Interventions: Device: Pulse CO-Oximeter Sensor

INTERVENTIONS:
Device: Pulse CO-Oximeter Sensor — Investigational Pulse CO-Oximeter sensor will measure hemoglobin (SpHb) and pleth variability index (PVi).
  Arms: Investigational Arm

SUMMARY:
This is a multicenter, cluster randomized controlled trial to assess the effects of an optimized intraoperative fluid and blood management strategy on postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of consent.
* Ability to provide written informed consent.
* Scheduled for non-urgent major surgery with general anesthesia
* At least one finger available and accessible for performing non-invasive pleth variability index (PVi) and hemoglobin (SpHb) monitoring.
* The Attending surgeon, attending anesthesiologist and the clinical care team agree with enrollment in the study, including the restrictions on monitoring procedures defined in the control group.

Exclusion Criteria:

* Untreated or uncontrolled hypertension defined as mean arterial pressure (MAP) greater than 120 mmHg, despite medications.
* Chronic kidney disease with glomerular filtration rate <30 ml/min/1.73 m2 or requiring renal-replacement therapy for end-stage renal disease.
* Surgeries where no bleeding is expected to occur (i.e., total knee surgery where blood loss is prevented by use of tourniquet).
* Surgeries performed in the prone position.
* Acute cardiovascular event, including acute or decompensated heart failure and acute coronary syndrome.
* Aortic pathology that could lead to misinterpretation of hemodynamic variables (e.g. intra- aortic balloon pump, thoracic aorta aneurysm).
* Renal vascular surgery.
* Preoperative sepsis.
* Circulatory shock.
* Preoperative vasoactive substance infusion before study entry.
* Concurrent participation in any interventional study.
* Pregnant or lactating women.
* Patients who refuse to receive blood transfusion(s).
* Patients with Do Not Resuscitate (DNR) orders.
* Open chest surgeries.
* Prisoners
* Patients for whom monitoring of CO, SV, PPV, and/or SVV to guide GDT or similar intra-operative fluid management, including continuous SpHb monitoring, would be standard of care.
* Patients have skin abnormalities affecting the digits such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown, nail polish or acrylic nails that would prevent the proper fit and application of the sensors.
* Cardio-pulmonary bypass (CPB) surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative complication | 7 days
  Occurrence of at least one post-operative complication by day 7 after surgery.